CLINICAL TRIAL: NCT00841217
Title: Effect of PPAR-Delta Agonist on Lipoprotein Kinetics in Metabolic Syndrome
Brief Title: Regulation of Lipoprotein Transport in Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Western Australia (Other)
Collaborators: National Heart Foundation, Australia (Other)
Responsible Party: Prof P Hugh R Barrett, University of Western Australia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UWA_PHR022009
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Obesity; Lipid Disorders; Cardiovascular Disease
Keywords: Drug treatment
MeSH Terms: conditions — Obesity; Lipid Metabolism Disorders; Cardiovascular Diseases | interventions — GW 501516

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo group
  Interventions: Drug: placebo pill
- 2 (Active Comparator): GW501516, 2.5mg
  Interventions: Drug: GW501516

INTERVENTIONS:
Drug: GW501516 — 2.5mg/day
  Arms: 2
Drug: placebo pill
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether PPAR-delta agonist (GW5015156)had favorable effect on lipoprotein metabolism.

DETAILED DESCRIPTION:
The metabolic syndrome (MetS) portends diabetes and cardiovascular disease (CVD). Dyslipoproteinaemia, reflected by elevated plasma triglyceride and reduced high-density lipoprotein (HDL) concentrations, is a cardinal feature of MetS that independently predicts CVD and is accordingly a therapeutic target for risk reduction. GW5015156 is a new PPAR-delta agonist that could be used to treat dyslipidemia in insulin resistance and obesity. However, the precise mechanisms of action of this agent on lipoprotein kinetics in MetS subjects have not yet fully been investigated. We therefore carried out a study to study the effect of GW5015156 on lipoprotein transport in subject with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Any three of the following:

  * Waist circumference > 102 cm
  * Triglycerides > 150 mg/dL
  * HDL-cholesterol < 40 mg/dL
  * Blood glucose > 110 mhg/dL
  * Blood pressures > 130/85 mmHg

Exclusion Criteria:

* Triglycerides > 500 mg/dL
* Diabetes mellitus
* CVD
* Consumption of > 30 g alcohol/day
* Use of agents affecting lipid metabolism
* APOE2/E2 genotype
* Creatinemia (> 120 umol/L)
* Hypothyroidism
* Abnormal liver and muscle enzymes

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-04; Primary Completion 2005-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
ApoB transport rate | 5 weeks

SECONDARY OUTCOMES:
ApoA and C-III transport rate | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Western Australia, Perth, Western Australia, Australia

REFERENCES:
- [Derived] Ooi EM, Watts GF, Sprecher DL, Chan DC, Barrett PH. Mechanism of action of a peroxisome proliferator-activated receptor (PPAR)-delta agonist on lipoprotein metabolism in dyslipidemic subjects with central obesity. J Clin Endocrinol Metab. 2011 Oct;96(10):E1568-76. doi: 10.1210/jc.2011-1131. Epub 2011 Aug 3. PMID 21816786